CLINICAL TRIAL: NCT07240051
Title: Assessment of the Efficacy and Safety of 50% Glycolic Acid, 30% Salicylic Acid, and Modified Jessner's Chemical Peels in the Treatment of Active Acne and Post-acne Hyperpigmentation: Randomized Controlled Trial
Brief Title: Efficacy of Different Types of Chemical Peels in the Treatment of Acne Vulgaris
Acronym: AV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nahla Maher Mahmoud Mahran (Other)
Responsible Party: Sponsor-Investigator, Nahla Maher Mahmoud Mahran, lecturer of Dermatology, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-327-2023
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acne; Peeling
Keywords: acne vulgaris; chemical peeling
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- glycolic acid group (Active Comparator): 30 patients received 50% glycolic acid peels
  Interventions: Procedure: Glycolic acid peel alone
- Salicylic acid group (Active Comparator): 30 patients received Salicylic acid 30%
  Interventions: Procedure: salicylic acid
- Modified Jessener group (Active Comparator): 30 patients received MJ peel
  Interventions: Procedure: modified jessener

INTERVENTIONS:
Procedure: Glycolic acid peel alone — Using a cotton tip applicator, a single coat of commercially prepared 50% GA peeling agent was evenly applied to the patient's face. Neutralization of the peel was done on reaching uniform erythema (endpoint) within 3-5 minutes. If frosting was observed in any area before the set time or endpoint, the area was neutralized with sodium bicarbonate
  Arms: glycolic acid group
Procedure: salicylic acid — Using a cotton tip applicator, a single coat of commercially prepared 30% SA peeling agent was evenly applied to the patient's face, moving from the forehead and advancing to the cheeks, chin, glabella, nose, and perioral area. Once white crystallization appeared, patients were asked to wash their faces with water.
  Arms: Salicylic acid group
Procedure: modified jessener — Commercially prepared MJ peel was applied using a gauze piece and light hand pressure. A single coat of peel was uniformly applied over the entire face. The coat was allowed to dry completely until erythema or frosting occurred, at which point patients were asked to wash their faces with cold water.
  Arms: Modified Jessener group

SUMMARY:
Assessment of the Efficacy and Safety of 50% Glycolic Acid, 30% Salicylic Acid, and Modified Jessner's Chemical Peels in the Treatment of Active Acne and Post-acne Hyperpigmentation: Randomized Controlled Trial.

ELIGIBILITY:
Inclusion Criteria:

* Facial active acne (mild and moderate cases)
* post-acne hyperpigmentation
* a minimum age of 18 years
* skin phototype III or IV

Exclusion Criteria:

* Pregnant or nursing women
* active infection in the treatment area (e.g., verrucae and herpes simplex)
* systemic disease (hypertension, diabetes, or bleeding tendency)
* systemic retinoid or laser treatment within the last 6 months
* history of keloidal tendency or Aspirin sensitivity.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
improvement in acne vulgaris by assessing Global acne scoring system and post-acne hyperpigmentation index | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No